CLINICAL TRIAL: NCT00593710
Title: A Randomized Double-blind Study Assessing the Effects of Losartan Versus Atenolol on Pulse Wave Velocity and the Biophysical Properties of the Aorta in Patients With Marfan Syndrome
Brief Title: Losartan Versus Atenolol for the Treatment of Marfan Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H07-01816
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Marfan Syndrome
Keywords: Randomized; double-blind superiority trial
MeSH Terms: conditions — Marfan Syndrome | interventions — Losartan; Atenolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Losartan
  Interventions: Drug: Losartan
- 2 (Active Comparator): Atenolol
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Losartan — Losartan (25mg OD)
  Arms: 1
Drug: Atenolol — Atenolol (25-50mg OD)
  Arms: 2

SUMMARY:
Marfan syndrome is a genetic disease of our connective tissue, which provides material and support for our skeleton, muscles, blood vessels and other parts of our bodies. People with Marfan syndrome may be tall and thin with slender, tapering fingers, long arms and legs, and spine curvature. They often have heart and eye problems. In some patients, the condition is very mild and the person has few or no symptoms. Others are always at risk of life-threatening problems, which usually involve damage to the valves in the heart or weakening of the large blood vessels leading from the heart. If the blood vessels become weak, they can balloon out (dilate) and break (rupture), which might cause the person to die suddenly. We have only a limited ability to stop the progression of disease in Marfan syndrome. Typically we use medicines that lower heart rate or blood pressure (or both). But this does not prevent the disease and very few drugs work well enough to keep patients from needing surgery or dying suddenly because a blood vessel has torn open. Our objective is to study two medicines to see if one, or both, can improve blood vessel function in patients with Marfan syndrome. One (Atenolol) belongs to a group of drugs called beta blockers and is often used to treat high blood pressure. It is the most common drug that is currently used to treat patients with Marfan syndrome. The other (Losartan) is also used for high blood pressure, but works in a different way. This study will help us to find better ways to treat people who have Marfan syndrome and to identify early changes in blood vessel function that may help to prevent long-term complications.

DETAILED DESCRIPTION:
The objective of the proposed research is to conduct a randomized, double-blind superiority feasibility study to compare the effects of two types of medication (Losartan, an Angiotensin Receptor Blocker, and Atenolol, a beta blocker) on vascular function in patients with Marfan syndrome (MFS). Our outcomes will include measuring the pulse wave velocity (PWV) and other biophysical properties of the aorta in the two groups of patients. This study will provide essential pilot data and development of logistics to enable a full multi-centre randomized controlled trial to test the hypothesis that Losartan will improve vascular function and, in the long-term, slow the rate of aortic root dilation.

MFS is an inherited disorder that affects 1:5000 of the population (i.e., 6000 people) in Canada alone. In MFS, mutations in the FBN1 gene lead to production of abnormal fibrillin 1 and to connective tissue abnormalities that impair skeletal, ocular, pulmonary and, most importantly, cardiovascular systems. Cardiovascular complications are also related to endothelial dysfunction, which has widespread implications for the health of large and muscular blood vessels and has effects on blood pressure, thrombosis, cholesterol levels and general vascular homeostasis. In MFS, progressive dilation, dissection and rupture of the aortic root may occur. This dilation is not solely due to the primary abnormality in collagen caused by the abnormal fibrillin protein. It remains unclear what the vascular mechanisms are that cause dilation of the aortic root. Eventual aortic rupture is a major cause of sudden death in MFS. If untreated, MFS significantly shortens the lifespan of affected individuals: half will succumb in their late 20s or early 30s, usually of aortic rupture. As such, it is crucial to develop effective treatments for cardiovascular disease in MFS and to improve our ability to detect critical changes in blood vessel (aortic) structure and function.

Clinical management of cardiovascular disease in individuals with MFS aims to decrease the rate of aortic root dilation and reduce the risk of dissection and rupture. Beta blockers (eg. Atenolol) have been the traditional medical treatment although some studies have cited the success of calcium antagonists or angiotensin converting enzyme (ACE) inhibitors, However, while beta blocker treatment has been successful in reducing the rate of dilation of the aorta, and its complications in MFS, studies report inconsistent responses to treatment and one pediatric study showed no benefit of beta blockers and better results with ACE inhibitors. Thus, it is still unclear whether one or the other of these pharmacological agents improves outcomes in regard to aortic dilation or rupture.

Recently, individuals with MFS have been shown to have dysregulation of transforming growth factor beta (TGF-beta) signaling that is postulated to result in the enlarged aortic root and other manifestations of the disease. Conversely, disorders of TGF beta 1 and 2 receptors have been shown to produce a Marfan phenotype. A study using a Marfan mouse model found that Losartan, an angiotensin 2 AT1 receptor blocker, prevented the development of aortic root dilation and other phenotypic manifestations of the syndrome. Among the actions of Losartan is the prevention of increased levels of TGF beta and its effects on stimulation of production of extracellular matrix in vascular smooth muscle. This evidence suggests that agents that alter TGF beta signalling, such as Losartan, might have significant potential to ameliorate endothelial dysfunction and aortic dilation in MFS. A clinical trial comparing the effects of Losartan with the current standard treatment regimen (beta blockers) is needed.

Ultimately, even treated individuals suffer from aortic dilation, so that surgical repair of the dilated aortic root is definitive in MFS. Elective surgery carries a low mortality and has significantly improved life expectancy; in contrast, emergency surgery for aortic root dissection or rupture carries a much higher mortality. Our earlier clinical studies and more recent work in a Marfan mouse model study suggest that aortic root dilation is a later stage in the disease process, which has involved cellular mechanisms (perhaps related to TGF beta) before aortic root dilation occurs. This suggests that, through research, one might enable clinicians to identify individuals who are in the early stages of vessel dilation and/or who are at risk for aortic rupture. If we could improve our capacity for early diagnosis of aortic root dilation, we could intervene in the pre-clinical stages and minimize the incidence of emergency surgery or sudden death.

Towards this goal, our group has developed a novel method of assessing the biophysical properties of the aorta by standard Echo Doppler techniques and have developed an accurate measure of PWV, which is considered the most important index of vascular function. In patients with MFS, we have demonstrated increased pulse wave velocity, reduced distensibility, increased stiffness in the large central arteries, and endothelial dysfunction-even if the aortic root had not yet dilated (see appended paper).

On the basis of these studies, we have also been given access to proprietary GE software to analyze raw data and have developed a software program that analyses the Doppler pulse flow and external carotid artery pressure tracing raw data to obtain parameters that previously required invasive techniques or laborious manual techniques to calculate. Using this new technique, which is unique to our group and applicable to other conditions that affect the aorta, we can now measure several key variables of aortic vessel function, including vascular distensibility, stiffness indices, impedances, total arterial compliance, reflective wave index, left ventricular work and efficiency. We predict that using this method to make a comprehensive assessment of aortic vascular (dys)function will provide for early detection of vascular changes and enable an improved comparison of the effectiveness of pharmacological treatment of cardiovascular disease in MFS.

Therefore, the objective of the proposed research is to use this methodology to compare aortic vascular function in individuals with MFS under conventional treatment using a beta blocker (Atenolol) or an angiotensin receptor blocker (Losartan). We propose a randomized, prospective, double-blinded superiority study to compare the actions of Losartan with Atenolol on vascular function in a group of 30 patients with MFS. Our research group has the unique capability to perform an analysis of the vascular effects of these therapies.

The Specific Aims are as follows:

1. To determine whether 12 months of treatment with Losartan decreases PWV more than 12 months of treatment with Atenolol in a cohort of patients with MFS;
2. To determine whether 12 months of treatment with Losartan will improve indices of distensibility, stiffness, arterial compliance, impedances and endothelial function more than 12 months of treatment with Atenolol in the same cohort of patients with MFS;
3. To determine whether 12 months of treatment with Losartan slows the progression of aortic root dilation when compared to 12 months of treatment with Atenolol in the same cohort of patients with MFS.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must conform to the diagnostic criteria for MFS;
2. Subjects must be between 12 and 25 years;
3. Subjects must have technically suitable echocardiographic windows to obtain the images needed to calculate the biophysical properties listed as outcome measures;
4. Subjects must provide informed consent and/or assent.

Exclusion Criteria:

1. Patients with significant aortic or mitral valve regurgitation;
2. Patients with a medical condition that would preclude them from taking either of the study medications or be taken off either medication for a brief period of time;
3. Female patients who are pregnant, planning to become pregnant, or breast-feeding.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2008-01; Primary Completion 2010-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pulse Wave Velocity | 12 months

SECONDARY OUTCOMES:
Biophysical properties of the aorta | 12 months
Brachial artery reactivity | 12 months
Aortic root dimension and area | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: George Sandor, MD, FRCPC, Principal Investigator — University of British Columbia; Cornelius van Breemen, MD, Study Director — University of British Columbia; James E. Potts, MD, Study Director — University of British Columbia
Locations (1):
- Children's Heart Centre, British Columbia's Children's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Sandor GG, Alghamdi MH, Raffin LA, Potts MT, Williams LD, Potts JE, Kiess M, van Breemen C. A randomized, double blind pilot study to assess the effects of losartan vs. atenolol on the biophysical properties of the aorta in patients with Marfan and Loeys-Dietz syndromes. Int J Cardiol. 2015 Jan 20;179:470-5. doi: 10.1016/j.ijcard.2014.11.082. Epub 2014 Nov 8. PMID 25465809